**PRODUCT:** Lofexidine granules for reconstitution (oral)

PROTOCOL NUMBER / AMENDMENT: USWM-LX2-1001 / 4

### **SPONSOR:**

USWM, LLC 4441 Springdale Rd. Louisville, KY 40241 United States of America (USA)

### TITLE:

A Study to Evaluate the Relative Bioavailability of a Test Formulation of Lofexidine Granules for Reconstitution and the Effect on Food on the Bioavailability of the Test Formula in Healthy Adult Subjects

**DOCUMENT DATE:** March 23, 2021

**IND NUMBER:** 47857

NCT NUMBER: NCT04188730

### STATISTICAL ANALYSIS PLAN

**STUDY TITLE** 

A study to evaluate the relative bioavailability of a test formulation of lofexidine granules for reconstitution and the effect of food on the bioavailability of the test formulation in healthy adult subjects

PROTOCOL NO.

USWM-LX2-1001 (Amendment 4)

SPONSOR USWM, LLC

4441 Springdale Rd. Louisville, KY 40241

United States of America (USA)

CLINICAL RESEARCH ORGANIZATION

DATE AND VERSION

23 Mar 2021 – Version 1.0 - Final

# **SAP Final Version Approvals**

A study to evaluate the relative bioavailability of a test formulation of lofexidine granules for reconstitution and the effect of food on the bioavailability of the test formulation in healthy adult subjects

| Written By: | Date: 24 Mur 2021 |
|-------------------------|-------------------|
| Reviewed By: | Date: 23 Man 2021 |
| Approved By: Signature: | Date: |

| STATISTICAL ANALYSIS PLAN | |
|------------------------------------------------------|----------------|
| PROTOCOL No. USWM-LX2-1001/ | |
| LOFEXIDINE GRANULES FOR RECONSTITUTION (ORAL) FORMUL | ATION, 90 uG/M |

# **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|-----------|-------------|-------------------------------|------------|
| Draft 0.1 | 19 Feb 2021 | New Document | |
| Draft 0.2 | 05 Mar 2021 | Incorporated Sponsor Comments | |
| Draft 0.3 | 18 Mar 2021 | Incorporated Sponsor Comments | |
| Final 1.0 | 23 Mar 2021 | Finalized Document | |

### **List of Abbreviations and Definition of Terms**

ADAE Analysis Dataset of Adverse Events
ADPC Analysis Dataset of PK Concentrations
ADPP Analysis Dataset of PK Parameters
ADSL Subject Level Analysis Dataset

AE Adverse Event

AUC $_{0-\infty}$  Area under the plasma concentration-time curve from time zero to

infinity

AUC<sub>0-t</sub> Area under the plasma concentration-time curve from time zero to

the time of last measurable concentration (t)

BMI Body Mass Index bpm Beats per minute

CL/F Apparent total clearance of the drug from plasma

C<sub>max</sub>
 C-SSRS
 Columbia-Suicide Severity Rating Scale
 C<sub>t</sub>
 Last measurable plasma concentration

CV Coefficient of variation ECG Electrocardiogram

eCRF Electronic Case Report Form

EQ Equivalent to

FDA Food and Drug Administration FSH Follicle Stimulating Hormone

g Gram hr Hour

ICH International Council for Harmonisation

in Inch

ISCV Intra-subject coefficient of variation

kg Kilogram

 $\lambda_z$  Apparent first-order terminal elimination rate constant

m<sup>2</sup> Meters squared Max. Maximum

Mean Arithmetic mean

MedDRA Medical Dictionary for Regulatory Activities

 $\begin{array}{ccc} mg & Milligram \\ \mu g & Microgram \\ min & Minute \\ Min. & Minimum \\ mL & Milliliter \end{array}$ 

mmHg Millimeter of mercury

msec Millisecond

PI Principal Investigator
PK Pharmacokinetic(s)
PR PR interval of the ECG
QRS QRS interval of the ECG

PROTOCOL No. USWM-LX2-1001 /

# Lofexidine Granules for Reconstitution (oral) Formulation, 90 µg/mL

| QT | QT interval of the ECG |
|-----|---------------------------|
| QTc | Corrected QT interval |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |

 $T_{1/2}$  First-order terminal elimination half-life TEAE Treatment Emergent Adverse Event

T<sub>max</sub> Time of maximum observed plasma concentration

 $V_Z/F$  Apparent volume of distribution during the terminal phase

## TABLE OF CONTENTS

| STATISTICAL ANALYSIS PLAN | 1 |
|---|---|
| SAP Final Version Approvals | 2 |
| Revision History | 3 |
| List of Abbreviations and Definition of Terms | 4 |
| TABLE OF CONTENTS | 6 |
| 1. INTRODUCTION | 9 |
| 2. STUDY OBJECTIVES | 9 |
| 3. OVERALL STUDY DESIGN | 9 |
| STUDY SCHEMATIC | 11 |
| 4. RANDOMIZATION | 12 |
| 5. SAMPLE SIZE | 12 |
| 6. ANALYSIS POPULATIONS | 12 |
| 6.1 Pharmacokinetic Population | 12 |
| 6.2 Safety Population | |
| 7. STATISTICAL ANALYSIS METHODS | 12 |
| 7.1 Baseline Characteristics | 13 |
| 7.1.1 Baseline Demographics | 13 |
| 7.1.2 Medical History | 13 |
| 7.2 Pharmacokinetic and Statistical Analyses | 13 |
| 7.2.1 Pharmacokinetic Parameters | |
| 7.2.2 Statistical Analyses | 14 |
| 7.3 Safety Analysis | |
| 7.3.1 Adverse Events | |
| 7.3.2 Vital Signs | 15 |
| 7.3.3 ECG | 15 |
| 7.3.4 Physical Examination | 16 |
| 7.3.5 Concomitant Medications | 16 |
| 7.3.6 Clinical Laboratory Tests | 16 |
| 7.3.7 C-SSRS Assessments | 16 |
| 7.4 Taste Assessment | 16 |
| 7.5 Multiple Comparisons | |
| 7.6 Interim Analyses | |
| 8. PK Reconciliation | |
| 9. TABLE, LISTING AND FIGURE SHELLS | |
| Table 10.1.1 Subject Disposition | |
| Table 11.2.1 Summary of Demographic Data (Safety Population) | 19 |
| Table 11.4.1.1 Summary of Pharmacokinetic Parameters of Untransformed Data: | |
| Lofexidine (N = XX subjects) | 20 |
| Table 11.4.1.2: Summary of Primary Endpoints Based on Plasma Lofexidine | |
| Concentrations (Ln-transformed): Treatment A vs. Treatment B (Fasted BE) | 22 |

| Table 11.4.1.3: Summary of Primary Endpoints Based on Plasma Lofexidine | |
|---|---|
| Concentrations (Ln-transformed): Treatment C vs. Treatment A (Food Effect) | 23 |
| Table 12.2.2.1 Summary of Treatment-Emergent Adverse Events by System Organ | |
| Class and MedDRA Preferred Term | 24 |
| Table 12.5.1 Summary of Vital Signs | 25 |
| Table 12.5.2 Shift Table for Changes from Baseline in ECGs | 26 |
| Table 12.5.3 Columbia-Suicide Severity Rating Scale – Ideation and Behavior | 27 |
| Table 12.5.4 Columbia-Suicide Severity Rating Scale – Most Severe Ideation | 28 |
| Table 14.2.1 Summary of Plasma Lofexidine Concentrations (units/mL) – (Treatment | |
| A) | 29 |
| Table 14.2.2 Summary of Plasma Lofexidine Concentrations (units/mL) – (Treatment | |
| B) | 29 |
| Table 14.2.3 Summary of Plasma Lofexidine Concentrations (units/mL) – (Treatment | |
| C) | 29 |
| Table 14.2.4 Summary of PK Parameters Based on Plasma Lofexidine Concentrations – | |
| (Treatment A) | 30 |
| Table 14.2.5 Summary of PK Parameters Based on Plasma Lofexidine Concentrations – | |
| (Treatment B) | 30 |
| Table 14.2.6 Summary of PK Parameters Based on Plasma Lofexidine Concentrations – | 2.0 |
| (Treatment C) | |
| Table 14.2.7 Summary of Taste Assessment Questionnaire Results (Treatment A or C) | |
| Listing 16.2.1 Discontinued Subjects. | |
| Listing 16.2.2 Protocol Deviations | |
| Listing 16.2.3 Subjects Excluded from Statistical Analysis | |
| Listing 16.2.4.1 Subject Demographics | |
| Listing 16.2.4.2 Prior and Concomitant Medications | |
| Listing 16.2.5.1 Dosing Date, Time, and Treatment Schedule | |
| Listing 16.2.5.2 Deviations from Scheduled Collection Times | |
| Listing 16.2.5.3 Taste Assessment Questionnaire (Treatment A or C) | |
| Listing 16.2.7 Adverse Events | |
| Listing 16.2.8.1 Serum Chemistry Laboratory Test Results | |
| Listing 16.2.8.2 Hematology Laboratory Test Results | |
| Listing 16.2.8.3 Urinalysis Laboratory Test Results | |
| Listing 16.2.8.4 Vital Signs | |
| Listing 16.2.8.5 Electrocardiogram Results | |
| Listing 16.2.8.6 Physical Examination Results | |
| Listing 16.2.8.7 Genotyping Results (If Applicable) | |
| Figure 11.4.1.1 Mean Plasma Lofexidine Concentrations | |
| Figure 11.4.1.2 Mean Plasma Lofexidine Concentrations – Semi-logarithmic Scale | 49 |
| Figure 14.2.1 Mean Plasma Lofexidine Concentrations (Including Error-bars) – | |
| Treatment A | 49 |

| Figure 14.2.2 Mean Plasma Lofexidine Concentrations (Including Error-bars) – | 40 |
|---|---|
| Treatment B. | 49 |
| Figure 14.2.3 Mean Plasma Lofexidine Concentrations (Including Error-bars) – | |
| Treatment C | 49 |
| Appendix 16.1.9 Individual Plasma Lofexidine Concentrations by Subject | 49 |
| Appendix 16.1.9 Individual Plasma Lofexidine Concentrations by Subject – Semi- | |
| logarithmic Scale | 49 |

| STATISTICAL ANALYSIS PLAN | | | | |
|---|---|---|---|---|
| PROTOCOL No. USWM-LX2-1001 / | | | | |
| LOFEXIDINE GRANULES FOR RECONSTITUTION | (ORAL | ) Formulation | ON, 90 μG | /MI |

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol USWM-LX2-1001 / Study No. (Amendment 4) dated 25 Jan 2021. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol USWM-LX2-1001 / Study No. (Amendment 4) dated 25 Jan 2021
- Note to File/Memo to File dated 08 Feb 2021
- Electronic Case Report Form (eCRF) Spec Version 1.1 dated 04 Mar 2021

This SAP has been developed and finalized prior to database lock of the clinical database for Protocol USWM-LX2-1001 / Study No.

#### 2. STUDY OBJECTIVES

The primary objectives of this study are:

- To evaluate the relative bioavailability of a test formulation of lofexidine granules for reconstitution (oral), final concentration 90 μg/mL (compared to the Orange Book RS/RLD product, LUCEMYRA tablets, EQ 0.18 mg base (US WorldMeds, LLC) under fasted conditions, and
- To evaluate the effect of food on the relative bioavailability of lofexidine granules for reconstitution (oral) when administered under fed compared to fasted conditions, following a single 0.36 mg dose to healthy adult male and female subjects.

The secondary objective is:

• To assess the safety and tolerability of a single 0.36 mg oral dose of lofexidine granules for reconstitution formulation when administered to healthy subjects under fasted and fed conditions.

#### 3. OVERALL STUDY DESIGN

This is an open-label, single-dose, randomized, three-treatment, three-period, four-sequence, crossover study comparing equal doses of the test formulation and reference product under fasted conditions and comparing the bioavailability of the granules for reconstitution (test formulation) under fed and fasted conditions. In two of the study periods, a single 0.36 mg dose of lofexidine will be administered to subjects following an overnight fast of at least 10 hours. In a third study period, a single 0.36 mg dose of lofexidine will be administered 30 minutes after the start of an

FDA-recommended standardized high-fat, high-calorie breakfast preceded by an overnight fast of at least 10 hours. The subjects will receive either lofexidine granules for reconstitution (oral)<sup>†</sup> (Treatment A or C) or two (2) LUCEMYRA tablets, EQ 0.18 mg base (Treatment B). The subjects will receive the test formulation in two of the study periods and the reference product in a third study period according to a four-sequence randomization schedule.

<sup>†</sup> The volume of lofexidine granules for reconstitution to be administered to subjects will be included in the Pharmacy Manual, to be provided by the Sponsor prior to study start.

Serial blood samples will be collected at pre-dose and at specified time points over 54 hours after dosing in each study period. Subjects will be confined at the clinical facility from at least 10.5 hours before dosing until after the 54-hour blood sample collection in each study period. The interval between doses will be at least 7 days.

The plasma concentrations of lofexidine will be measured by fully validated analytical procedures. Statistical analysis using an average bioavailability approach will be performed to estimate the bioavailability of the test formulation relative to the reference product under fasted conditions. The bioavailability of the granules for reconstitution (test formulation) under fasted and fed conditions will also be compared.

For evaluation of the safety endpoint, the following assessments will be performed throughout the study: collection of medical history and Adverse Events (AEs), laboratory tests, vital signs, physical examination, 12-lead electrocardiograms (ECGs), and Columbia Suicidality Severity Rating Scale (C-SSRS) assessments. No formal statistical testing will be performed on safety variables.

#### **STUDY SCHEMATIC**

| Study Phase | Screening | Perio | ds I, II | and I | II | End of Study |
|---|---|---|---|---|---|---|
| Activity | Within 28 days | Check-In | Day | Day | Day | Day 3 |
| Activity | of Day 1 | Day -1 | 1 | 2 | 3 | Period III |
| Informed Consent | X | | | | | |
| Social, Medical History and Demographic Data | X | | | | | |
| Physical Examination <sup>1</sup> | X | X | | | X | X |
| C-SSRS <sup>2</sup> | | X | | | X | X |
| Virology Testing | X | | | | | |
| FSH testing (if applicable) <sup>3</sup> | X | | | | | |
| 12 Lead ECG <sup>4</sup> | X | X | X | | X | X |
| Clinical Lab Tests <sup>5</sup> | X | | | | | X |
| Inclusion/Exclusion | X | | | | | |
| Eligibility | | X | | | | |
| Vital Signs <sup>4</sup> | X | X | X | | X | X |
| Drug and Alcohol Screen <sup>6</sup> | X | X | | | | |
| Serum Pregnancy Test <sup>7</sup> | X | | | | | X |
| Urine Pregnancy Test <sup>7</sup> | | X | | | | |
| Prior and Concomitant Medication | X | X | X | X | X | X |
| Confinement <sup>8</sup> | | X | X | X | X | |
| Genotype sampling <sup>9</sup> | | | X | | | |
| High-fat, high-calorie breakfast <sup>10</sup> | | | X | | | |
| Dosing <sup>11</sup> | | | X | | | |
| Taste Assessment <sup>12</sup> | | | X | | | |
| PK sampling <sup>13</sup> | | | X | X | X | |
| Adverse Events <sup>14</sup> | | X | X | X | X | X |

- 1. To be performed as specified in Sections 5.3.1.1 (screening) and 5.5.5 of the Clinical Study Protocol.
- 2. C-SSRS to be obtained as specified in Section 5.5.5 of the Clinical Study Protocol.
- 3. To be performed as specified in Appendix 8.1.6 of the Clinical Study Protocol, if applicable.
- 4. ECGs and vital signs to be measured as specified in Sections 5.3.1.1 and 5.3.3 (screening) and 5.5.5 of the Clinical Study Protocol. Note: ECG to be conducted at check-in for Periods II and III only.
- 5. Clinical laboratory tests (see Appendix 8.1.1 of the Clinical Study Protocol) to be performed as specified in Sections 5.3.1.1 (screening) and 5.5.4 of the Clinical Study Protocol.
- 6. For all subjects, test results must be negative before drug will be administered to the subject. Alcohol tested at check-in only. Drug and alcohol tests, as appropriate, to be performed as specified in Appendix 8.1.3 of the Clinical Study Protocol (at screening) and Appendix 8.1.4 of the Clinical Study Protocol (at check-in).
- 7. Female subjects only. For all female subjects, test results must be negative before drug will be administered to the subject. Pregnancy tests to be performed as specified in Appendix 8.1.5 of the Clinical Study Protocol.
- 8. Subjects should enter the clinical facility at least 10.5 hours before dosing and will remain confined until at least 54 hours after dosing in each study period.
- 9. Blood sample to be collected in Period I as specified in Appendix 8.1.2 of the Clinical Study Protocol.
- 10. The standardized high-fat, high-calorie breakfast will be provided as specified in Section 5.4.4 of the Clinical Study Protocol.
- 11. Single dose to be administered as specified in Section 5.4.1 of the Clinical Study Protocol.
- 12. Treatments A or C only. To be performed as outlined in Section 5.4.1 and Appendix 8.2 of the Clinical Study Protocol.
- 13. Blood samples to be collected as specified in Section 5.6 of the Clinical Study Protocol.
- 14. From dosing in Period I until the end of the study.

#### 4. RANDOMIZATION

Treatments will be administered according to a three-treatment, three-period, four-sequence design as outlined below. The randomization will be generated in blocks of four with each sequence occurring once in each block.

| Sequence | Period I | Period II | Period III |
|---|---|---|---|
| 1 (N=4) | Treatment B | Treatment A | Treatment C |
| 2 (N=4) | Treatment B | Treatment C | Treatment A |
| 3 (N=4) | Treatment A | Treatment C | Treatment B |
| 4 (N=4) | Treatment C | Treatment A | Treatment B |
| Treatment A = Lofexidine granules – fasted conditions | | | |
| Treatment B = LUCEMYRA tablets – fasted conditions | | | |
| Treatment C = Lofexidine granules – fed conditions | | | |

The randomization schedule will be generated by the Biostatistics Department at before the first dosing period using SAS®, Version 9.4 or higher.

### 5. SAMPLE SIZE

A sample size of 16 subjects enrolled to complete 12 subjects is considered, by the Sponsor, sufficient to meet the objectives of this study. The sample size for this study was determined based on clinical and practical considerations and not on a formal statistical power calculation.

#### 6. ANALYSIS POPULATIONS

### 6.1 Pharmacokinetic Population

Data from subjects who have sufficient plasma concentrations to characterize  $C_{max}$  and  $AUC_{0-t}$  of at least one of the study treatments (A, B or C) will be included in the pharmacokinetic analysis. Data from any subject/period that does not provide sufficient plasma concentrations to characterize  $C_{max}$  and  $AUC_{0-t}$  will be excluded from the pharmacokinetic analysis.

Data from subjects who have sufficient plasma concentrations to characterize  $C_{max}$  and  $AUC_{0-t}$  from at least two periods of the study, one of which includes Treatment A, will be included in the comparative statistical analysis.

### **6.2 Safety Population**

The safety population will include all subjects who are administered at least one dose of a study treatment (A, B or C).

#### 7. STATISTICAL ANALYSIS METHODS

Data will be summarized with respect to demographic, baseline characteristics, safety, and pharmacokinetic (PK) variables.

For categorical variables, the number and percent of each category within a parameter will be calculated for non-missing data. For continuous variables, statistics will include number of observations, mean, standard deviation, median, minimum, and maximum values.

#### 7.1 Baseline Characteristics

### 7.1.1 Baseline Demographics

Demographic information collected at screening includes age, sex, ethnicity, race, body weight (lbs), height (in), BMI, and tobacco use. Body weight and height will be converted into kg and cm, respectively, for presentation in listings and tables.

All data will be listed by subject. A summary table will be presented for the safety population.

### 7.1.2 Medical History

Only clinically significant medical history data, if they exist, will be presented and listed by subject.

### 7.2 Pharmacokinetic and Statistical Analyses

Pharmacokinetic and statistical services will be performed by SAS®, Version 9.4 or higher will be used for all pharmacokinetic and statistical calculations.

No concentration estimates will be provided for missing sample values. Any sample with a missing value will be treated as if the sample had not been scheduled for collection. Data from subjects with missing concentration values (such as missing blood draws, lost samples, samples unable to be quantified) may be used if pharmacokinetic parameters can be estimated using the remaining data points, otherwise data from these subjects will be excluded from the final analysis.

Descriptive statistics (n, mean, SD, % coefficient of variation [%CV], minimum, median, maximum, geometric mean, geometric CV) will be reported for lofexidine concentrations at each time point by treatment.

Linear and semi-logarithmic graphs of the concentration-time profiles for each subject will be provided, using the actual times of sample collections. Graphical presentations of mean results will use the scheduled times of sample collections. Actual sample collection time will be used for calculating the pharmacokinetic parameters, although data will be summarized referencing the scheduled sample collection times.

#### 7.2.1 Pharmacokinetic Parameters

The pharmacokinetic parameters will be determined from the plasma concentration data using a non-compartmental model.

For the test and reference products, the peak exposure  $(C_{max})$  will be the observed maximum plasma concentration; the time to peak exposure  $(T_{max})$  will be the collection time at which  $C_{max}$  is first observed.

Areas under the plasma concentration-time curve from time zero to the time of last measurable concentration (AUC<sub>0-t</sub>) will be calculated by the linear trapezoidal method. Area under the plasma concentration-time curve from time zero to time infinity (AUC<sub>0- $\infty$ </sub>) will be calculated as follows:

 $AUC_{0-\infty} = AUC_{0-t} + C_t/\lambda_z$ , where  $C_t$  is the last measurable plasma concentration and  $\lambda_z$  is the

apparent first-order terminal rate constant.

 $\lambda_z$  will be estimated, when possible, from the negative of the slope of the dataset with the best-fit least-squares linear regression analysis of the terminal ln-linear concentration-time data. The number of data points (3 or more) in the terminal phase (not including  $C_{max}$ ) to be included in the final regression analysis for an evaluable  $\lambda_z$  will be determined from the dataset that has the highest adjusted R-squared ( $R^2$ ) value of 0.7 or more.

 $\lambda_z$  will be considered non-evaluable if (1) the last three terminal points are used to determine  $\lambda_z$  and either the middle or the last point is higher than the preceding point or (2) the resulting adjusted  $R^2$  value is less than 0.7. An evaluable  $\lambda_z$  will be considered not reliable and not reportable if the resulting apparent first-order terminal half-life ( $T_{\frac{1}{2}}$ ) value is longer than the time interval over which  $\lambda_z$  is determined, an interval that is longer than the estimated  $T_{\frac{1}{2}}$  will be explored. The interval with the next highest adjusted  $R^2$  value will be chosen and the decrease in the adjusted  $R^2$  value will be assessed to determine if a reliable estimation of the  $\lambda_z$  is possible. If  $\lambda_z$  is deemed not reliable then no  $T_{\frac{1}{2}}$  and  $AUC_{0-\infty}$  values will be reported for that dataset.  $T_{\frac{1}{2}}$  will be calculated as  $\ln(2)/\lambda_z$ .

Apparent volume of distribution during the terminal phase  $(V_Z/F)$  of the drug from plasma will be calculated as follows: Dose /  $[AUC_{0-\infty} \cdot \lambda_Z]$ ).

Apparent total clearance of the drug from plasma (CL/F) will be calculated as follows: Dose /  $AUC_{0-\infty}$ .

Descriptive statistics (n, mean, SD, % coefficient of variation (%CV), geometric mean, minimum, median, maximum) will be reported for all PK parameters.

### 7.2.2 Statistical Analyses

A linear mixed effect model with treatment, sequence and period as fixed effects and random effects of subject nested within sequence will be used. Sequence effects will be tested against the Type III mean square term for subject-within sequence at the two-sided  $\alpha = 10\%$  level of significance. Least squares means for the treatments (LSMEANS statement), the differences between adjusted treatment means, and the standard errors associated with these differences (ESTIMATE statement) will be estimated.

Two-sided confidence intervals (90%) on the geometric mean ratios (obtained from logarithmic transformed data) for  $AUC_{0-t}$ ,  $AUC_{0-\infty}$  and  $C_{max}$  for the comparison of Treatment A to Treatment B (to compare the test formulation and reference product under fasted conditions) and the comparison of Treatment C to Treatment A (to compare the granules for reconstitution [test formulation] under fed and fasted conditions) will be constructed to test two one-sided hypotheses at the  $\alpha=0.05$  level of significance.

The statistical model will be conducted separately for Treatment A versus Treatment B analysis and for Treatment C versus Treatment A analysis using an incomplete block design.

#### 7.3 Safety Analysis

No formal statistical testing will be performed on safety variables.

#### 7.3.1 Adverse Events

Adverse events (AEs) and Serious Adverse Events (SAEs) will be collected through both solicited and unsolicited means from dosing in Period I until the end of the study.

All reported AEs will be coded and classified according to the MedDRA Version 23.0 or higher adverse event dictionary. Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship to study treatment, action taken and outcome. The severity is characterized as mild, moderate or severe. The relationship to the study treatment is characterized as unrelated or related.

Adverse events will be listed by subject, treatment, system organ class, and preferred term. The incidence of AEs will be summarized by system organ class (SOC), preferred term (PT) and treatment. Subjects will be counted once per preferred term and once per system organ class, per treatment. The system organ classes will be ordered by decreasing total frequency then alphabetically. The preferred terms within each system organ class will be ordered by decreasing total frequency then alphabetically.

The summary table for Adverse Events will be based upon the safety population. AEs and SAEs will be summarized by overall number of AEs in the final report text, per treatment. The number of AEs leading to withdrawal from the study or SAEs will also be summarized in text.

### 7.3.2 Vital Signs

Sitting/supine vital signs assessment (temperature, respiration rate, pulse, and blood pressure) and orthostatic blood pressure assessment (within 3 minutes of standing from a sitting/supine position) will be performed at the screening visit. Vital signs (temperature, pulse, and blood pressure) will be measured in the sitting position at check-in of each study period.

Blood pressure and pulse (sitting) will be measured at pre-dose (between -1.5 and -0.5 hours before dosing), and 3.5 and 7.5 hours ( $\pm$  30 minutes) after dosing in each study period and before release from the clinical facility in Periods I and II.

Descriptive statistics will be used to summarize the observed values by treatment at each time point and the change from baseline at each post-dose time point. Vital signs will be listed by subject.

#### 7.3.3 ECG

A 12-lead ECG will be conducted in triplicate for all subjects at the screening visit. A 12-lead ECG will also be performed at pre-dose (in triplicate) in Periods I, II and III (Day 1, before vital sign assessments) and 3.5 hours post-dose (± 30 minutes), at release from the clinic (Periods I and II), at check-in (Day -1) for Periods II and III, and at the end of the study (i.e., release from the clinic in Period III or early termination).

Safety (12-lead) ECG changes from baseline will be presented in a shift table (i.e., normal to abnormal) at each post-dose time point. Safety 12-lead ECG parameters will be listed by subject with any out of normal range values flagged.

### 7.3.4 Physical Examination

A complete physical examination (including height and weight) will be performed at screening. A brief physical examination will be performed at check-in of each study period and before release from the clinical facility in Periods I and II. At the end of the study (or early termination), all subjects will have a complete physical examination (including weight [NOT height]) performed.

Physical examination results will be listed by subject.

#### 7.3.5 Concomitant Medications

All prior and concomitant medications taken since screening until the end of the study will be listed by subject.

### 7.3.6 Clinical Laboratory Tests

All subjects will have chemistry, hematology, and urinalysis performed at screening and end of study.

Clinical laboratory results will be listed by subject and any clinically significant out of range laboratory results will be flagged.

#### 7.3.7 C-SSRS Assessments

Subjects will complete the Columbia Suicidality Severity Rating Scale (C-SSRS) at check-in for each study period, at release from the clinical facility in Periods I and II, and at the end of study (i.e., release from the clinical facility in Period III or early termination). The C-SSRS: Baseline document should be used at check-in for Period I and the C-SSRS: Since Last Visit document should be used in all other instances.

For categorical variables for C-SSRS data, the number and percent of each category within a parameter will be calculated for non-missing data and tabulated by time point.

#### 7.4 Taste Assessment

Within 10 minutes after completion of the dosing procedure for the subject's first dose of lofexidine granules (Treatment A or C), each subject will be required to complete a Taste Assessment Questionnaire.

Taste Assessment Questionnaire results will be listed by treatment then by subject.

### 7.5 Multiple Comparisons

No multiple comparison adjustment will be made in this study.

### 7.6 Interim Analyses

There is no interim analysis planned in this study.

#### 8. PK Reconciliation

Biostatistics team will reconcile the plasma concentration data sent by the bioanalytical laboratory

| STATISTICAL ANALYSIS PLAN | |
|---------------------------------|---------------------------------------|
| PROTOCOL No. USWM-LX2-1001 / | |
| LOFEXIDINE GRANULES FOR RECONST | ΓΙΤUTION (ORAL) FORMULATION, 90 μG/MI |

and the PK sample collection times from the SDTM dataset (i.e., BE domain). This reconcile step will be verified and documented appropriately.

### 9. TABLE, LISTING AND FIGURE SHELLS

The following shells are presented in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings, and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. In addition to the standard SDTM datasets; the ADaM datasets; ADSL, ADAE, ADPC and ADPP will be programmed and submitted.

# **Table 10.1.1 Subject Disposition**

| Subject Disposition | Overall<br>N = xx |
|-------------------------------------------------|-------------------|
| Subjects Randomized | xx (xx.x%) |
| Subjects included in Safety Population | xx (xx.x%) |
| Subjects included in Pharmacokinetic Population | xx (xx.x%) |
| Total Discontinued | xx (xx.x%) |
| Reason for Discontinuation | xx (xx.x%) |
| Adverse Event | xx (xx.x%) |
| Non-Compliance | xx (xx.x%) |
| Positive Substance Abuse Screen | xx (xx.x%) |
| Withdrawal by Subject | xx (xx.x%) |
| | xx (xx.x%) |

**Table 11.2.1 Summary of Demographic Data (Safety Population)** 

| | | Overall |
|----------------|-------------------------------------------|-----------------|
| | | N = xx |
| Age (years) | Mean ± SD | $xx.x \pm xx.x$ |
| | Range (Min., Max.) | XX, XX |
| | Median | XX |
| Age Groups | < 18 | x (xx.x%) |
| | 18 – 40 | x (xx.x%) |
| | 41 – 64 | x (xx.x%) |
| | 65 – 75 | x (xx.x%) |
| | > 75 | x (xx.x%) |
| Sex | Male | x (xx.x%) |
| | Female | x (xx.x%) |
| Ethnicity* | Hispanic or Latino | x (xx.x%) |
| | Not Hispanic or Latino | x (xx.x%) |
| Race* | American Indian or Alaska Native | x (xx.x%) |
| | Asian | x (xx.x%) |
| | Black or African American | x (xx.x%) |
| | Native Hawaiian or Other Pacific Islander | x (xx.x%) |
| | White | x (xx.x%) |
| | Multiple | x (xx.x%) |
| BMI | Mean ± SD | $xx.x \pm xx.x$ |
| $(kg/m^2)$ | Range (Min., Max.) | XX, XX |
| | Median | XX |
| Other Factors | | |
| Height | $Mean \pm SD$ | $xx.x \pm xx.x$ |
| (cm) | Range (Min., Max.) | XX, XX |
| | Median | XX |
| Weight | $Mean \pm SD$ | $xx.x \pm xx.x$ |
| (kg) | Range (Min., Max.) | XX, XX |
| | Median | XX |
| Tobacco Users† | Yes | x (xx.x%) |
| | No | x (xx.x%) |

<sup>\*</sup> Categories based on FDA Guidance "Collection of Race and Ethnicity Data in Clinical Trials", Issue Date: October 26, 2016.

<sup>†</sup> Defined as current tobacco user (having used tobacco- or nicotine-containing products within 30 days before initial dosing).

Table 11.4.1.1 Summary of Pharmacokinetic Parameters of Untransformed Data: Lofexidine (N = XX subjects)

| Pharmacokinetic<br>Parameter | Treatment | N<br>(# datasets) | Arithmetic mean ± SD<br>(%CV)* | Min. | Median | Max. |
|---|---|---|---|---|---|---|
| AUC <sub>0-t</sub><br>(units·hr/mL) | A | X | $\begin{aligned} xxx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | xxx.xxxx | xxx.xxxx | xxx.xxxx |
| | В | Х | $ \begin{array}{c} xxx.xxxx \pm xx.xxxx \\ (xx.xxxx) \end{array} $ | xxx.xxxx | XXX.XXXX | xxx.xxxx |
| | С | Х | $ \begin{aligned} xx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | xx.xxxx | XX.XXXX | xx.xxxx |
| AUC <sub>0-∞</sub><br>(units·hr/mL) | | | | xxx.xxxx | XXX.XXXX | xxx.xxxx |
| | B x xxx.xxxx ± xx.xxxx (xx.xxxx) | | xxx.xxxx | XXX.XXXX | xxx.xxxx | |
| | C x xx.xxxx ± xx.xxxx (xx.xxxx) | | xx.xxxx | XX.XXXX | xx.xxxx | |
| AUC <sub>0-t</sub> /<br>AUC <sub>0-∞</sub> | A | Х | $\begin{aligned} xxx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | xxx.xxxx | XXX.XXXX | xxx.xxxx |
| | В | Х | $\begin{aligned} xxx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | xxx.xxxx | XXX.XXXX | XXX.XXXX |
| | С | X | $ \begin{aligned} xx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | XX.XXXX | XX.XXXX | xx.xxxx |
| C <sub>max</sub><br>(units/mL) | A | Х | $\begin{aligned} xxx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | xxx.xxxx | XXX.XXXX | xxx.xxxx |
| | В | Х | $\begin{aligned} xxx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | xxx.xxxx | XXX.XXXX | xxx.xxxx |
| | С | X | $ \begin{aligned} xx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | XX.XXXX | XX.XXXX | xx.xxxx |
| T <sub>max</sub> (hr) | A | Х | $\begin{aligned} xxx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | xxx.xxxx | XXX.XXXX | xxx.xxxx |
| | В | X | $\begin{aligned} xxx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | xxx.xxxx | XXX.XXXX | XXX.XXXX |
| | С | Х | $ \begin{array}{c} xx.xxxx \pm xx.xxxx \\ (xx.xxxx) \end{array} $ | xx.xxxx | xx.xxxx | xx.xxxx |
| λ <sub>z</sub><br>(hr <sup>-1</sup> ) | A | Х | $ \begin{array}{c} xx.xxxx \pm xx.xxxx \\ (xx.xxxx) \end{array} $ | xx.xxxx | xx.xxxx | xx.xxxx |
| | В | Х | xx.xxxx ± xx.xxxx<br>(xx.xxxx) | xx.xxxx | xx.xxxx | xx.xxxx |
| | С | Х | $ \begin{aligned} xx.xxxx &\pm xx.xxxx \\ (xx.xxxx) \end{aligned}$ | XX.XXXX | XX.XXXX | xx.xxxx |

# Lofexidine Granules for Reconstitution (oral) Formulation, $90~\mu\text{G/mL}$

| Pharmacokinetic<br>Parameter | Treatment | N<br>(# datasets) | Arithmetic mean ± SD<br>(%CV)* | Min. | Median | Max. |
|---|---|---|---|---|---|---|
| T <sub>1/2</sub> (hr) | A | Х | $ \begin{array}{c} xx.xxxx \pm xx.xxxx \\ (xx.xxxx) \end{array} $ | xx.xxxx | xx.xxxx | XX.XXXX |
| | В | Х | $xx.xxxx \pm xx.xxxx$ $(xx.xxxx)$ | XX.XXXX | xx.xxxx | xx.xxxx |
| | С | X | xx.xxxx ± xx.xxxx<br>(xx.xxxx) | xx.xxxx | xx.xxxx | xx.xxxx |
| CL/F<br>(units) | A | X | $ xx.xxxx \pm xx.xxxx \\ (xx.xxxx)$ | xx.xxxx | xx.xxxx | xx.xxxx |
| | В | Х | $xx.xxxx \pm xx.xxxx (xx.xxxx)$ | xx.xxxx | xx.xxxx | xx.xxxx |
| | С | X | $ xx.xxxx \pm xx.xxxx \\ (xx.xxxx)$ | xx.xxxx | xx.xxxx | xx.xxxx |
| V <sub>z</sub> /F (units) | A | Х | $xx.xxxx \pm xx.xxxx (xx.xxxx)$ | xx.xxxx | xx.xxxx | xx.xxxx |
| | В | Х | $ xx.xxxx \pm xx.xxxx \\ (xx.xxxx)$ | xx.xxxx | xx.xxxx | xx.xxxx |
| | С | Х | $ \begin{array}{c} xx.xxxx \pm xx.xxxx \\ (xx.xxxx) \end{array} $ | xx.xxxx | XX.XXXX | xx.xxxx |

<sup>\* %</sup>CV is calculated as 100\*SD/Mean

Table 11.4.1.2: Summary of Primary Endpoints Based on Plasma Lofexidine Concentrations (Ln-transformed): Treatment A vs. Treatment B (Fasted BE)

| Parameter | Trt. | LS<br>Geometric<br>Mean | Standard<br>Error | Geometric CV | Contrast<br>(# subjects) | LSGM<br>Ratio<br>(%) | 90%<br>Confidence<br>Interval (%) | ISCV (%)* | P-value<br>Period | P-value<br>Sequence | 90% CI<br>within 80-<br>125% |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AUC <sub>0-t</sub> (units·hr/mL) | A | XX | XX | xx.x | A vs B $(n = xx)$ | XX. XX | xx. xx - xx. xx | xx.x | x.xxxx | x.xxxx | Yes/No |
| | В | XX | XX | XX.X | | | | | | | |
| AUC₀-∞<br>(units·hr /mL) | A | xx | XX | XX.X | A vs B $(n = xx)$ | xx. xx | xx. xx - xx. xx | xx.x | x.xxxx | x.xxxx | Yes/No |
| | В | XX | XX | xx.x | | | | | | | |
| C <sub>max</sub> (units/mL) | A | XX | XX | XX.X | A vs B $(n = xx)$ | xx. xx | xx. xx - xx. xx | xx.x | x.xxxx | x.xxxx | Yes/No |
| | В | xx | XX | xx.x | | | | | | | |

<sup>\*</sup> ISCV (Intra-subject coefficient of variation) is calculated as sqrt[exp(MSE)-1] using the model mean square error.

Table 11.4.1.3: Summary of Primary Endpoints Based on Plasma Lofexidine Concentrations (Ln-transformed): Treatment C vs. Treatment A (Food Effect)

| Parameter | Trt. | LS<br>Geometric<br>Mean | Standard<br>Error | Geometric CV | Contrast<br>(# subjects) | LSGM<br>Ratio<br>(%) | 90%<br>Confidence<br>Interval (%) | ISCV (%)* | P-value<br>Period | P-value<br>Sequence | 90% CI<br>within 80-<br>125% |
|---|---|---|---|---|---|---|---|---|---|---|---|
| AUC <sub>0-t</sub> (units·hr/mL) | С | XX | XX | xx.x | C vs A $(n = xx)$ | xx. xx | xx. xx - xx. xx | xx.x | x.xxxx | x.xxxx | Yes/No |
| | A | XX | XX | XX.X | | | | | | | |
| AUC <sub>0-∞</sub> (units·hr /mL) | С | xx | XX | XX.X | C vs A $(n = xx)$ | xx. xx | xx. xx - xx. xx | xx.x | x.xxxx | x.xxxx | Yes/No |
| | A | XX | XX | xx.x | | | | | | | |
| C <sub>max</sub> (units/mL) | С | XX | XX | XX.X | C vs A $(n = xx)$ | xx. xx | xx. xx - xx. xx | xx.x | x.xxxx | x.xxxx | Yes/No |
| | A | xx | XX | xx.x | | | | | | | |

<sup>\*</sup> ISCV is calculated as sqrt[exp(MSE)-1] using the model mean square error.

LOFEXIDINE GRANULES FOR RECONSTITUTION (ORAL) FORMULATION, 90 µG/ML

Table 12.2.2.1 Summary of Treatment-Emergent Adverse Events by System Organ Class and MedDRA Preferred Term

| System Organ Class/MedDRA Preferred Term | Treatment A<br>n (%) | Treatment B<br>n (%) | Treatment C<br>n (%) | Overall<br>n (%) |
|---|---|---|---|---|
| Subjects having at least one TEAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| System Organ Class | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Preferred Term | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

Subjects counted once per preferred term and once per system organ class, per treatment.

Treatment A = ## subjects dosed.

Treatment B = ## subjects dosed.

Treatment C = ## subjects dosed.

Page 1 of N Created on: DDMMMYYYY

Programming Note 1: Subjects with more than one PT for the same SOC will be counted only once. Subjects with more than one incidence of same PT will be counted only once.

Programming Note 2: The system organ classes will be ordered by decreasing overall frequency then alphabetically. The preferred terms within each system organ class will be ordered by decreasing overall frequency then alphabetically

n = Number of subjects reporting AE

<sup>% = (</sup>Number of subjects reporting AE / number of subjects dosed with respective study drug) x 100

**Table 12.5.1 Summary of Vital Signs** 

| | | | | Obser | rved Data | | | Change f | rom Baseli | ne |
|---|---|---|---|---|---|---|---|---|---|---|
| Evaluation | Treatment | Time Point | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| Diastolic<br>Blood | A | Pre-dose<br>(Baseline) | XX | xx.x (xx.x) | xx.x | xx.x, xx.x | | | | |
| Pressure | A | 3.5 hr | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | XX | xx.x (xx.x) | xx.x | xx.x, xx.x |
| (mmHg) | A | 7.5 hr | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | XX | xx.x (xx.x) | XX.X | xx.x, xx.x |
| | | etc. | | | | | | | | |
| | В | Pre-dose<br>(Baseline) | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | | | | |
| | В | 3.5 hr | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | XX | xx.x (xx.x) | XX.X | xx.x, xx.x |
| | В | 7.5 hr | XX | xx.x(xx.x) | XX.X | xx.x, xx.x | XX | xx.x(xx.x) | XX.X | xx.x, xx.x |
| | | etc. | | | | | | | | |
| | С | Pre-dose<br>(Baseline) | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | | | | |
| | C | 3.5 hr | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | XX | xx.x (xx.x) | XX.X | xx.x, xx.x |
| | C | 7.5 hr | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | XX | xx.x (xx.x) | XX.X | xx.x, xx.x |
| | | etc. | | | | | | | | |
| Pulse (beats/min) | A | Pre-dose<br>(Baseline) | XX | xx.x (xx.x) | xx.x | xx.x, xx.x | | | | |
| | A | 3.5 hr | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | XX | xx.x (xx.x) | xx.x | xx.x, xx.x |
| | A | 7.5 hr | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | XX | xx.x (xx.x) | xx.x | xx.x, xx.x |
| | | etc. | | | | | | | | |


Programming Note: If any pre-dose assessment data are missing, the nearest non-missing pre-dose value will be used as the baseline.

**Table 12.5.2 Shift Table for Changes from Baseline in ECGs** 

| | | 3.5 | Hours Post- | dose | | Release | |
|---|---|---|---|---|---|---|---|
| Treatment | Pre-dose<br>(Baseline) | Normal<br>n (%) | Abnormal (NCS) n (%) | Abnormal<br>(CS)<br>n (%) | Normal<br>n (%) | Abnormal (NCS) n (%) | Abnormal<br>(CS)<br>n (%) |
| A | Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Abnormal (NCS) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Abnormal (CS) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| В | Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Abnormal (NCS) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Abnormal (CS) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | ••• | | | | | | |

Created on: DDMMMYYYY

Page 1 of N

Table 12.5.3 Columbia-Suicide Severity Rating Scale – Ideation and Behavior

| C-SSRS Question | Period I<br>Check-in –<br>Lifetime<br>n (%) | Period I<br>Release –<br>Since Last Visit<br>n (%) | Period II<br>Check-in –<br>Since Last Visit<br>n (%) | Period II<br>Release –<br>Since Last Visit<br>n (%) | Period III<br>Check-in –<br>Since Last Visit<br>n (%) | Period III<br>Release/Early<br>Termination –<br>Since Last Visit<br>n (%) |
|---|---|---|---|---|---|---|
| Suicidal Ideation | | | | | | |
| Wish to be dead | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Non-specific active suicidal thoughts | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Active suicidal ideation with any methods (not plan) without intent to act | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Active suicidal ideation with some intent to act, without specific plan | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Active suicidal ideation with specific plan and intent | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Suicidal Behavior | | | | | | |
| Engaged in non-suicidal self-injurious behavior | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Preparatory acts or behavior | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Suicidal behavior | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Actual attempt | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Interrupted attempt | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Aborted attempt | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Suicide | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

n = Number of subjects who experience the event (i.e., respond 'Yes')

<sup>%</sup> = (Number of subjects who experience the event / number of subjects dosed) x 100

**Table 12.5.4 Columbia-Suicide Severity Rating Scale – Most Severe Ideation** 

| C-SSRS Question | Visit | 1<br>n (%) | 2<br>n (%) | 3<br>n (%) | 4<br>n (%) | 5<br>n (%) | 0<br>n (%) |
|---|---|---|---|---|---|---|---|
| Most severe ideation type no. | Period I Check-in – Lifetime | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Frequency | Period I Check-in – Lifetime | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Duration | Period I Check-in – Lifetime | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Controllability | Period I Check-in – Lifetime | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Deterrents | Period I Check-in – Lifetime | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Reasons for ideation | Period I Check-in – Lifetime | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Most severe ideation type no. | Period I Release – Since Last Visit | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Frequency | Period I Release – Since Last Visit | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ••• | | | | | | | |

 $<sup>\</sup>overline{n}$  = Number of subjects in category % = (Number of subjects in category / number of subjects dosed) × 100

LOFEXIDINE GRANULES FOR RECONSTITUTION (ORAL) FORMULATION, 90 µG/ML

Table 14.2.1 Summary of Plasma Lofexidine Concentrations (units/mL) – (Treatment A)

| Sub. | Per. | Seq. | Pre-<br>dose | 0.5<br>hr | 0.75<br>hr | 1.0<br>hr | 1.5<br>hr | 2.0<br>hr | 3.0<br>hr | 4.0<br>hr | 5.0<br>hr | 7.0<br>hr | 10.0<br>hr | 16.0<br>hr | 24.0<br>hr | 30.0<br>hr | <br>54.0<br>hr |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 3001 | | | | | | | | | | | | | | | | | |
| | X | X | X.XX | X.XX | X.XX | | | | | | | | | | | | |
| 3002 | X | X | X.XX | X.XX | X.XX | | | | | | | | | | | | |
| 3003 | X | X | X.XX | X.XX | x.xx | etc. | | | | | | | | | | | |
| 3004 | X | X | X.XX | x.xx | x.xx | | | | | | | | | | | | |
| 3005 | X | X | x.xx | x.xx | x.xx | | | | | | | | | | | | |
| ••• | | | | | | | | | | | | | | | | | |
| 3.7 | 1 1 | | | 1 | 1 | 1 | 1 | | 1 | 1 | | 1 | 1 | 1 | 1 | 1 | |
| N | | | | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | | | | |
| St. Dev. | | | | | | | | | | | | | | | | | |
| CV (%) | | | | | | | | | | | | | | | | | |
| Min. | | | | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | | | | |
| Max. | | | | | | | | | | | | | | | | | |
| Geometric<br>Mean | | | | | | | | | | | | | | | | | |
| Geometric<br>CV (%) | | | | | | | | | | | | | | | | | |


Note: Similar listings will be produced for Treatment B and Treatment C.

Table 14.2.2 Summary of Plasma Lofexidine Concentrations (units/mL) – (Treatment B)

Table 14.2.3 Summary of Plasma Lofexidine Concentrations (units/mL) – (Treatment C)

Table 14.2.4 Summary of PK Parameters Based on Plasma Lofexidine Concentrations – (Treatment A)

| Sub. | Per. | Seq. | AUC 0-t<br>(units·hr/mL) | AUC 0-∞<br>(units·hr/mL) | AUC 0-t/<br>AUC0-∞ | C <sub>max</sub> (units/mL) | T <sub>max</sub> (h) | λ <sub>z</sub> (hr <sup>-1</sup> ) | T <sub>1/2</sub> (hr) | CL/F<br>(units) | V <sub>z</sub> /F<br>(units) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 3001 | Х | х | X.XXX | x.xxx | x.xxx | x.xxxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx |
| 3002 | Х | х | X.XXX | x.xxx | x.xxx | x.xxxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx |
| 3003 | Х | Х | X.XXX | x.xxx | x.xxx | x.xxxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx |
| 3004 | Х | Х | X.XXX | x.xxx | X.XXX | x.xxxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx |
| 3005 | X | X | X.XXX | x.xxx | x.xxx | x.xxxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx |
| N | | | | | | | | | | | |
| N | | | | | | | | | | | |
| Mean | | | | | | | | | | | |
| St. Dev. | | | | | | | | | | | |
| CV (%) | | | | | | | | | | | |
| Min. | | | | | | | | | | | |
| Median | | | | | | | | | | | |
| Max. | | | | | | | | | | | |
| Geometric Mean | | | | | | | | | | | |
| Geometric CV (%) | | | | | | | | | | | |


Note: A similar table will be produced for Treatment B and Treatment C.

Table 14.2.5 Summary of PK Parameters Based on Plasma Lofexidine Concentrations – (Treatment B)

Table 14.2.6 Summary of PK Parameters Based on Plasma Lofexidine Concentrations – (Treatment C)

Table 14.2.7 Summary of Taste Assessment Questionnaire Results (Treatment A or C)

| | Treatment A N = xx n (%) | Treatment C $N = xx$ $n (\%)$ |
|---|---|---|
| Overall Taste | | |
| Like very much | x (xx.x%) | x (xx.x%) |
| Like moderately | x (xx.x%) | x (xx.x%) |
| Like slightly | x (xx.x%) | x (xx.x%) |
| Neither like nor dislike | x (xx.x%) | x (xx.x%) |
| Dislike slightly | x (xx.x%) | x (xx.x%) |
| Dislike moderately | x (xx.x%) | x (xx.x%) |
| Dislike very much | x (xx.x%) | x (xx.x%) |
| Sourness | | |
| Like very much | x (xx.x%) | x (xx.x%) |
| Like moderately | x (xx.x%) | x (xx.x%) |
| Like slightly | x (xx.x%) | x (xx.x%) |
| Neither like nor dislike | x (xx.x%) | x (xx.x%) |
| Dislike slightly | x (xx.x%) | x (xx.x%) |
| Dislike moderately | x (xx.x%) | x (xx.x%) |
| Dislike very much | x (xx.x%) | x (xx.x%) |
| Bitterness | | |
| Like very much | x (xx.x%) | x (xx.x%) |
| Like moderately | x (xx.x%) | x (xx.x%) |
| Like slightly | x (xx.x%) | x (xx.x%) |
| Neither like nor dislike | x (xx.x%) | x (xx.x%) |
| Dislike slightly | x (xx.x%) | x (xx.x%) |

# LOFEXIDINE GRANULES FOR RECONSTITUTION (ORAL) FORMULATION, 90 μG/ML

| | Treatment A | Treatment C |
|--------------------------|-------------|-------------|
| | N = xx | N = xx |
| | n (%) | n (%) |
| Dislike moderately | x (xx.x%) | x (xx.x%) |
| Dislike very much | x (xx.x%) | x (xx.x%) |
| Mouthfeel/Texture | | |
| Like very much | x (xx.x%) | x (xx.x%) |
| Like moderately | x (xx.x%) | x (xx.x%) |
| Like slightly | x (xx.x%) | x (xx.x%) |
| Neither like nor dislike | x (xx.x%) | x (xx.x%) |
| Dislike slightly | x (xx.x%) | x (xx.x%) |
| Dislike moderately | x (xx.x%) | x (xx.x%) |
| Dislike very much | x (xx.x%) | x (xx.x%) |
| Grittiness | | |
| Like very much | x (xx.x%) | x (xx.x%) |
| Like moderately | x (xx.x%) | x (xx.x%) |
| Like slightly | x (xx.x%) | x (xx.x%) |
| Neither like nor dislike | x (xx.x%) | x (xx.x%) |
| Dislike slightly | x (xx.x%) | x (xx.x%) |
| Dislike moderately | x (xx.x%) | x (xx.x%) |
| Dislike very much | x (xx.x%) | x (xx.x%) |
| Aftertaste | | |
| Like very much | x (xx.x%) | x (xx.x%) |
| Like moderately | x (xx.x%) | x (xx.x%) |
| Like slightly | x (xx.x%) | x (xx.x%) |
| Neither like nor dislike | x (xx.x%) | x (xx.x%) |

# LOFEXIDINE GRANULES FOR RECONSTITUTION (ORAL) FORMULATION, 90 μG/ML

| | Treatment A N = xx n (%) | Treatment C N = xx n (%) |
|--------------------|----------------------------|--------------------------|
| Dislike slightly | x (xx.x%) | x (xx.x%) |
| Dislike moderately | x (xx.x%) | x (xx.x%) |
| Dislike very much | x (xx.x%) | x (xx.x%) |

# **Listing 16.2.1 Discontinued Subjects**

| Subject<br>No. | Discontinuation Reason | Date of<br>Discontinuation | Time of<br>Discontinuation | Discontinuation<br>Related to COVID-19<br>Pandemic |
|---|---|---|---|---|
| XXXX | Withdrawal By Subject | dd/Mmm/yyyy | hh:mm | |
| XXXX | Withdrawal By Subject | dd/Mmm/yyyy | hh:mm | |


Programming Notes: Listings will be presented by subject number. Secondary fields for AEs, PDs, and Other must be listed

# **Listing 16.2.2 Protocol Deviations**

| Subject No. | Type of Protocol Deviation | Deviation Date | PD Related to<br>COVID-19 Pandemic |
|---|---|---|---|
| XXXX | Consumption or use of a restricted item | dd/Mmm/yyyy | |
| XXXX | Assessment performed out of window: Vital signs | dd/Mmm/yyyy | |
| ••• | | | |


Programming Note: Secondary fields for deviation categories of Assessment Not Performed and Assessment Performed Out of Window are required to be presented.
**Listing 16.2.3 Subjects Excluded from Statistical Analysis** 

| Sub. | Excluded from Analysis | Reason for Exclusion from Analysis | Applicable Treatment(s) |
|---|---|---|---|
| XXXX | A vs B | Subject did not have sufficient pharmacokinetic data for this analysis | В |
| XXXX | A vs B , C vs A | Pre-dose concentration > 5% of C <sub>max</sub> | A |
| XXXX | C vs A | C <sub>max</sub> observed at first post-dose sampling timepoint | C |
| XXXX | A vs B, C vs A | Data excluded because of protocol deviation | B, C |

# **Listing 16.2.4.1 Subject Demographics**

| Subject<br>No. | Sex | Age<br>(yrs) | Ethnicity | Race | Tobacco<br>User | Height (in) | Weight (lbs) | BMI (kg/m²) |
|---|---|---|---|---|---|---|---|---|
| XXXX | Male | 43 | Not Hispanic or Latino | Black or African American | No | XX | XX | XX.X |
| xxxx | Male | 36 | Not Hispanic or Latino | Black or African American | No | xx | XX | xx.x |

#### **Listing 16.2.4.2 Prior and Concomitant Medications**

| Subject<br>No. | Medication | Indication | Dose | Route | Frequency* | Date Started | Date Stopped | Therapeutic<br>Drug Class |
|---|---|---|---|---|---|---|---|---|
| XXXX | Vitamin D | General health | 1000 IU | Oral | QD | /Mmm/yyyy | Ongoing | |
| XXXX | Multivitamin | General health | 1 Tablet | Oral | QD | dd/Mmm/yyyy | dd/Mmm/yyyy | |

<sup>\*</sup>PRN - As needed; QD - Daily (once per day); Q4H - Every 4 hours; Q8H - Every 8 hours; Q12H - Every 12 hours; BID - Twice per day; TID - 3 times per day; QID - 4 times per day; QOD - Every other day; QS - Every week; QM - Every month; Q3M - Every 3 months


Programming Note: Only the applicable abbreviations need to be included in the footnote.

LOFEXIDINE GRANULES FOR RECONSTITUTION (ORAL) FORMULATION, 90 µG/ML

Listing 16.2.5.1 Dosing Date, Time, and Treatment Schedule

| Subject No. | Period | Date | Time | Treatment |
|-------------|--------|-------------|-------|-----------|
| xxxx | I | dd/Mmm/yyyy | hh:mm | A |
| xxxx | II | dd/Mmm/yyyy | hh:mm | В |
| xxxx | III | dd/Mmm/yyyy | hh:mm | C |
| xxxx | I | dd/Mmm/yyyy | hh:mm | C |
| xxxx | II | dd/Mmm/yyyy | hh:mm | A |
| xxxx | III | dd/Mmm/yyyy | hh:mm | В |
| xxxx | I | dd/Mmm/yyyy | hh:mm | В |
| xxxx | II | dd/Mmm/yyyy | hh:mm | A |
| xxxx | III | dd/Mmm/yyyy | hh:mm | C |

Page 1 of N Created on: DDMMMYYYY

**Listing 16.2.5.2 Deviations from Scheduled Collection Times** 

| Subject No. | Treatment | Period | Sample Time (hrs) | Deviation* |
|-------------|-----------|--------|----------------------|------------|
| xxxx | A | I | 10.0 | +3 |
| xxxx | В | II | $0.5-54.0^{\dagger}$ | DFP |
| XXXX | C | III | 5.0 | +4 |
| xxxx | В | I | 16.0 | +3 |
| xxxx | A | II | 48.0 | NS |

<sup>\*</sup> Minutes assessment was performed late (+) or early (-).

DFP: Dropped from Period DFS: Dropped from Study NS: No Sample Collected

<sup>†</sup>Subject did not participate in this portion of the study

**Listing 16.2.5.3 Taste Assessment Questionnaire (Treatment A or C)** 

| Subject<br>No. | Treatment* | Overall Taste | Smell | Sweetness | Sourness | Bitterness | Mouthfeel/<br>Texture | Grittiness | Aftertaste |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | A | Like very much | Like very much | Like very much | Like very much | Like very much | Like very much | Like very much | Like very much |
| XXXX | A | Like<br>moderately | Like<br>moderately | Like<br>moderately | Like<br>moderately | Like<br>moderately | Like<br>moderately | Like<br>moderately | Like<br>moderately |
| xxxx | A | Like slightly | Like slightly | Like slightly | Like slightly | Like slightly | Like slightly | Like slightly | Like slightly |
| XXXX | A | Neither like nor dislike | Neither like nor dislike | Neither like nor<br>dislike | Neither like nor dislike | Neither like nor dislike | Neither like nor dislike | Neither like nor dislike | Neither like nor dislike |
| xxxx | С | Dislike slightly | Dislike slightly | Dislike slightly | Dislike slightly | Dislike slightly | Dislike slightly | Dislike slightly | Dislike slightly |
| xxxx | С | Dislike<br>moderately | Dislike<br>moderately | Dislike<br>moderately | Dislike<br>moderately | Dislike<br>moderately | Dislike<br>moderately | Dislike<br>moderately | Dislike<br>moderately |
| xxxx | С | Dislike very much | Dislike very much | Dislike very much | Dislike very much | Dislike very much | Dislike very much | Dislike very much | Dislike very much |
| | | | 1 . 1 | | | | 1: | | |

<sup>\*</sup>Taste Assessment Questionnaire completed once by each subject, only after the subject's first dose of lofexidine granules (Treatment A or C).

## **Listing 16.2.7 Adverse Events**

| Subject<br>No. | System Organ Class/<br>MedDRA Preferred Term/<br>AE Term | Treatment | Onset<br>Date<br>Time | Onset<br>Date<br>Time | Severity | Relationship | Outcome | Action<br>Taken<br>with Study<br>Treatment | Other<br>Action<br>Taken | SAE |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | Nervous system disorders /<br>Headache / Headache | A | dd/Mmm/yyyy<br>hh:mm | dd/Mmm/yyyy<br>hh:mm | Mild | Unrelated | Recovered/<br>Resolved | Dose Not<br>Changed | None | No |
| XXXX | Investigations / Blood<br>pressure increased / Blood<br>pressure increased | С | dd/Mmm/yyyy<br>hh:mm | dd/Mmm/yyyy<br>hh:mm | Moderate | Related | Recovered/<br>Resolved | Dose Not<br>Changed | None | No |
| ••• | | | | | | | | | | |

**Listing 16.2.8.1 Serum Chemistry Laboratory Test Results** 

| Subject<br>No. | Visit | Date | Time | Test | Result | Units | Clinically Significant (if out of range) |
|---|---|---|---|---|---|---|---|
| XXXX | Screening | dd/Mmm/yyyy | hh:mm | Alanine Aminotransferase | XX.X | U/L | |
| XXXX | Screening | dd/Mmm/yyyy | hh:mm | Alkaline Phosphatase | XX.X | U/L | |
| XXXX | Screening | dd/Mmm/yyyy | hh:mm | Aspartate Aminotransferase | XX.X | U/L | |
| xxxx | Screening | dd/Mmm/yyyy | hh:mm | Bilirubin | XX.X | mg/dL | |
| XXXX | Screening | dd/Mmm/yyyy | hh:mm | Creatinine | XX.X | mg/dL | |
| XXXX | Screening | dd/Mmm/yyyy | hh:mm | Glucose | XX.X | mg/dL | |
| xxxx | Screening | dd/Mmm/yyyy | hh:mm | Potassium | XX.X | mmol/L | |
| xxxx | Screening | dd/Mmm/yyyy | hh:mm | Urea Nitrogen | XX.X | mg/dL | |
| XXXX | Screening | dd/Mmm/yyyy | hh:mm | Magnesium | XX.X | mg/dL | |
| XXXX | Screening | dd/Mmm/yyyy | hh:mm | Sodium | XX.X | mEq/L | |
| XXXX | Screening | dd/Mmm/yyyy | hh:mm | Chloride | XX.X | mEq/L | |
| xxxx | End of Study/<br>Early Termination | dd/Mmm/yyyy | hh:mm | Alanine Aminotransferase | XX.X | U/L | |

Note: Similar listings will be produced for hematology and urinalysis.

#### **Listing 16.2.8.2 Hematology Laboratory Test Results**

### **Listing 16.2.8.3 Urinalysis Laboratory Test Results**

#### **Listing 16.2.8.4 Vital Signs**

| Subject<br>No. | Treatment | Visit | Time Point | Date | Time | Vital Sign | Result | Units | Clinically<br>Significant<br>(if out of<br>range) |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | | Screening | | dd/Mmm/yyyy | hh:mm | Diastolic Blood Pressure | XX | mmHg | |
| XXXX | | Screening | | dd/Mmm/yyyy | hh:mm | Pulse | XX | beats/min | |
| XXXX | | Screening | | dd/Mmm/yyyy | hh:mm | Respiration Rate | XX | breaths/min | |
| XXXX | | Screening | | dd/Mmm/yyyy | hh:mm | Systolic Blood Pressure | XXX | mmHg | |
| XXXX | | Screening | | dd/Mmm/yyyy | hh:mm | Temperature | XX.X | F | |
| XXXX | | Screening Repeat 1 | | dd/Mmm/yyyy | hh:mm | Diastolic Blood Pressure | XX | mmHg | |
| XXXX | | Screening Repeat 1 | | dd/Mmm/yyyy | hh:mm | Systolic Blood Pressure | XXX | mmHg | |
| XXXX | A | Period I | Check-in | dd/Mmm/yyyy | hh:mm | Diastolic Blood Pressure | XX | mmHg | |
| XXXX | A | Period I | Check-in | dd/Mmm/yyyy | hh:mm | Pulse | XX | beats/min | |
| XXXX | A | Period I | Check-in | dd/Mmm/yyyy | hh:mm | Systolic Blood Pressure | XXX | mmHg | |
| XXXX | A | Period I | Check-in | dd/Mmm/yyyy | hh:mm | Temperature | XX.X | F | |
| XXXX | A | Period I | Pre-dose | dd/Mmm/yyyy | hh:mm | Diastolic Blood Pressure | XX | mmHg | |
| XXXX | A | Period I | Pre-dose | dd/Mmm/yyyy | hh:mm | Pulse | XX | beats/min | |
| XXXX | A | Period I | Pre-dose | dd/Mmm/yyyy | hh:mm | Systolic Blood Pressure | XXX | mmHg | |
| XXXX | A | Period I | 3.5 hr | dd/Mmm/yyyy | hh:mm | Diastolic Blood Pressure | XX | mmHg | |
| XXXX | A | Period I | 3.5 hr | dd/Mmm/yyyy | hh:mm | Pulse | XX | beats/min | |
| XXXX | A | Period I | 3.5 hr | dd/Mmm/yyyy | hh:mm | Systolic Blood Pressure | XXX | mmHg | |
| XXXX | A | Period I | 7.5 hr | dd/Mmm/yyyy | hh:mm | Diastolic Blood Pressure | XX | mmHg | |
| | | | ••• | | | | | | |

**Listing 16.2.8.5 Electrocardiogram Results** 

| | | | | | | | Intervals (msec) | | | ec) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>No. | Treatment | Visit | Time Point | Date | Time | Vent.<br>Rate<br>(bpm) | PR | QRS | QT | QTc | Result | Clinical<br>Significance<br>(if abnormal) |
| xxxx | | Screening | | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | | Screening | | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | | Screening | | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | A | Period I | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | A | Period I | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | A | Period I | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | A | Period I | 3.5 hr | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | A | Period I | Release | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | | Period II | Check-in | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | | Period II | Check-in | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | xxx | Normal<br>Variant | |
| xxxx | | Period II | Check-in | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | В | Period II | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | xxx | Normal | |
| xxxx | В | Period II | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | В | Period II | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | В | Period II | 3.5 hr | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | xxx | Abnormal | Clinically<br>Significant |
| xxxx | В | Period II | Release | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | | Period III | Check-in | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | | Period III | Check-in | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | | Period III | Check-in | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | C | Period III | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | C | Period III | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | C | Period III | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| xxxx | C | Period III | 3.5 hr | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |

| | | | | | | | Intervals (msec) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>No. | Treatment | Visit | Time Point | Date | Time | Vent.<br>Rate<br>(bpm) | PR | QRS | QT | QTc | Result | Clinical<br>Significance<br>(if abnormal) |
| xxxx | С | Period III | Release | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | xxx | XXX | Abnormal | Not Clinically<br>Significant |
| xxxx | | Screening | | dd/Mmm/yyyy | hh:mm | XX | xxx | xxx | xxx | xxx | Normal | |
| XXXX | В | Period I | Pre-dose | dd/Mmm/yyyy | hh:mm | XX | XXX | XXX | XXX | XXX | Normal | |
| ••• | | | | | | | | | | | | |

**Listing 16.2.8.6 Physical Examination Results** 

| Subject<br>No. | Treatment | Visit | Time Point | Category | Result | Description (if abnormal/changed) |
|---|---|---|---|---|---|---|
| xxxx | | | | General Appearance | | |
| XXXX | | Screening | | Skin | Abnormal | |
| XXXX | | Screening | | EENT | | |
| XXXX | | Screening | | Head | | |
| XXXX | | Screening | | Neurological | | |
| XXXX | | Screening | | Cardiovascular | | |
| XXXX | | Screening | | Lungs/Thorax | | |
| XXXX | | Screening | | Abdominal | | |
| XXXX | | Screening | | Musculoskeletal | | |
| XXXX | | Screening | | Extremities | | |
| xxxx | A | Period I | Check-in | General Appearance | No Change | |
| XXXX | A | Period I | Check-in | Cardiovascular | Change | |
| XXXX | A | Period I | Check-in | Lungs/Thorax | | |
| XXXX | A | Period I | Check-in | Abdominal | | |
| XXXX | A | Period I | Release | General Appearance | | |
| xxxx | A | Period I | Release | Cardiovascular | | |
| XXXX | A | Period I | Release | Lungs/Thorax | | |
| XXXX | A | Period I | Release | Abdominal | | |
| XXXX | В | Period II | Check-in | General Appearance | | |

## **Listing 16.2.8.7 Genotyping Results (If Applicable)**

| Subject No. | CYP2D6 Metabolizer Status |
|-------------|---------------------------|
| xxxx | Extensive Metabolizer |
| XXXX | Intermediate Metabolizer |
| XXXX | Poor Metabolizer |
| XXXX | Ultrarapid Metabolizer |

Figure 11.4.1.1 Mean Plasma Lofexidine Concentrations

Figure 11.4.1.2 Mean Plasma Lofexidine Concentrations – Semi-logarithmic Scale

Figure 14.2.1 Mean Plasma Lofexidine Concentrations (Including Error-bars) – Treatment A

Figure 14.2.2 Mean Plasma Lofexidine Concentrations (Including Error-bars) – Treatment B

Figure 14.2.3 Mean Plasma Lofexidine Concentrations (Including Error-bars) – Treatment C

Appendix 16.1.9 Individual Plasma Lofexidine Concentrations by Subject

Appendix 16.1.9 Individual Plasma Lofexidine Concentrations by Subject – Semi-logarithmic Scale